CLINICAL TRIAL: NCT00033111
Title: Phase 2, Double-Blind, Placebo Controlled Trial of Cabergoline for the Treatment of Cocaine Dependence
Brief Title: A Study of Cabergoline for the Treatment of Cocaine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-CTO-0007-1; NCT00024895 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabergoline (Active Comparator): Subjects received one tablet of 0.5 mg of cabergoline tablet per week for 12 weeks.
  Interventions: Drug: Cabergoline
- Placebo (Placebo Comparator): Subjects received one tablet of 0.5 mg of cabergoline matched placebo tablet per week for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cabergoline
  Other Names: Dostinex
  Arms: Cabergoline
Drug: Placebo — sugar pill manufactured to mimic cabergoline 05mg tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess cabergoline for the Treatment of Cocaine Dependence

DETAILED DESCRIPTION:
To assess the efficacy and safety of cabergoline in reducing cocaine use in subjects with cocaine dependence. This is a DB, placebo-controlled, parallel group design study where subjects will receive either .5mg cabergoline or placebo for 12 weeks with a 4 week follow-up.

ELIGIBILITY:
Inclusion Criteria:

Must have a DSM-4 criteria for cocaine dependence; be seeking treatment for cocaine dependence; have the ability to understand and provide written informed consent; females of child-bearing potential using proper method of birth control.

Exclusion Criteria:

Additional criteria available during screening at the site.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2001-06; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of cabergoline in reducing cocaine use in subjects with cocaine dependence | Week 12
  Success in the reduction of cocaine use was determined by comparing cocaine non-use days (self-report confirmed or disproved by urine BE level at each study visit) expressed as the weekly mean proportion of non-use days to the total number of non-missing study days that week.

SECONDARY OUTCOMES:
Reduction in cocaine use | 12 weeks
  Measured by the weekly mean proportion of non-use days according to the subject's self report without regard to BE levels

CONTACTS AND LOCATIONS:
Overall Officials: Steve Shoptaw, Ph.D., Principal Investigator — Friends Research Institute, Inc.
Locations (2):
- United States (2):
  - Torrance Clinic, Torrance, California
  - Medical University of South Carolina, Charleston, South Carolina